CLINICAL TRIAL: NCT01967576
Title: Phase II Study of Axitinib (AG-013736) With Evaluation of the VEGF-pathway in Metastatic, Recurrent or Primary Unresectable Pheochromocytoma/Paraganglioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Apolo, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140001; 14-C-0001
Record Dates: First submitted 2013-10-19; First posted 2013-10-23 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Mutation in SDHB gene; Mutation in SDHV gene; Mutation in VHL gene; Pharmacogenomics analyses; Germline DNA examination
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1-Axitinib (Experimental): Axitinib 5 mg twice a day on a 28-day cycle
  Interventions: Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Axitinib (AG-013736) — 5 mg twice a day on a 28-day cycle.
  Other Names: INLYTA

SUMMARY:
Background:

* Most treatments for malignant pheochromocytomas/paragangliomas (PHEO/PGL) are palliative and multidisciplinary. Chemotherapy using the combination of cyclophosphamide, vincristine, and dacarbazine has been successfully utilized in the management of rapidly progressive metastatic PHEO, with more than 50% complete or partial tumor response and more than 70% complete or partial biochemical response.
* Vascular endothelial growth factor (VEGF) expression and evidence of angiogenesis has been found in many PHEO/PGL, so it is plausible that interfering with VEGF signaling may result in anti-tumor activity in patients with PHEO/PGL.
* Axitinib (AG-013736) is an oral, potent and selective inhibitor of vascular endothelial growth factor (VEGF) receptors 1, 2, and 3. Pre-clinical data suggests that the anti-tumor activity of axitinib may result from its anti-angiogenic activity and that this is reversible when treatment is discontinued.
* Given the known clinical safety and efficacy of axitinib, an assessment of its activity in PHEO/PGL and its impact on the VEGF pathway in PHEO/PGL could provide valuable information.

Objectives:

* Determine the response rate of metastatic PHEO/PGL to axitinib (AG-013736).
* Determine the progression-free survival of metastatic PHEO/PGL treated with axitinib (AG-013736).
* Explore the relationship of potential biological markers of axitinib activity with clinical outcomes.
* Perform pharmacogenomics analyses of drug metabolism and transport proteins through germline deoxyribonucleic acid (DNA) examination.

Eligibility:

* Adults with a confirmed pathologic diagnosis of PHEO/PGL by the Laboratory of Pathology, National Cancer Institute (NCI)
* Biochemical evidence of PHEO/PGL
* Imaging confirmation of metastatic, locally advanced or unresectable disease.
* Measurable disease at presentation
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Patients must not have received prior therapy with a tyrosine kinase (TK) inhibitor

Design:

* Phase II, open label, non-randomized trial
* Patients with metastatic pheochromocytoma/paraganglioma will receive axitinib (AG-013736 twice a day (BID)) in eight-week cycles
* Patients will be evaluated for response every eight weeks using Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Tumor biopsies are not mandatory but every attempt will be made to obtain these from patients prior to starting axitinib and again 20 - 30 days after treatment has begun.
* Approximately 12 to 37 patients will be needed to achieve the objectives of the trial

DETAILED DESCRIPTION:
Background:

* Most treatments for malignant pheochromocytomas/paragangliomas (PHEO/PGL) are palliative and multidisciplinary. Chemotherapy using the combination of cyclophosphamide, vincristine, and dacarbazine has been successfully utilized in the management of rapidly progressive metastatic PHEO, with more than 50% complete or partial tumor response and more than 70% complete or partial biochemical response.
* Vascular endothelial growth factor (VEGF) expression and evidence of angiogenesis has been found in many PHEO/PGL, so it is plausible that interfering with VEGF signaling may result in anti-tumor activity in patients with PHEO/PGL.
* Axitinib (AG-013736) is an oral, potent and selective inhibitor of vascular endothelial growth factor (VEGF) receptors 1, 2, and 3. Pre-clinical data suggests that the anti-tumor activity of axitinib may result from its anti-angiogenic activity and that this is reversible when treatment is discontinued.
* Given the known clinical safety and efficacy of axitinib, an assessment of its activity in PHEO/PGL and its impact on the VEGF pathway in PHEO/PGL could provide valuable information.

Objectives:

* Determine the response rate of metastatic PHEO/PGL to axitinib (AG-013736).
* Determine the progression-free survival of metastatic PHEO/PGL treated with axitinib (AG-013736).
* Explore the relationship of potential biological markers of axitinib activity with clinical outcomes.
* Perform pharmacogenomics analyses of drug metabolism and transport proteins through germline deoxyribonucleic acid (DNA) examination.

Eligibility:

* Adults with a confirmed pathologic diagnosis of PHEO/PGL by the Laboratory of Pathology, National Cancer Institute (NCI)
* Biochemical evidence of PHEO/PGL
* Imaging confirmation of metastatic, locally advanced or unresectable disease.
* Measurable disease at presentation
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Patients must not have received prior therapy with a tyrosine kinase (TK) inhibitor

Design:

* Phase II, open label, non-randomized trial
* Patients with metastatic pheochromocytoma/paraganglioma will receive axitinib (AG-013736 twice a day (BID)) in eight-week cycles
* Patients will be evaluated for response every twelve weeks (+/- 1 week) using Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Approximately 12 to 37 patients will be needed to achieve the objectives of the trial

ELIGIBILITY:
* INCLUSION CRITERIA

2.1.1 Adults with a confirmed pathologic diagnosis of pheochromocytoma/paraganglioma by the Laboratory of Pathology, National Cancer Institute (NCI) when such tissue is available to confirm or

In the event that outside tissue is not available:

* an outside pathology report confirms the diagnosis of Pheo-PGI, AND
* the patient has nuclear medicine imaging studies that would only be positive in an adult patient with a diagnosis of Pheo/PGL (Fluorodopa (F-DOPA), Dotatate, F-Dopamine or Metaiodobenzylguanidine (MIBG))

2.1.1.1 Imaging confirmation of metastatic disease

2.1.1.2 Measurable disease at the time of enrollment per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

2.1.1.3 A life expectancy of at least 3 months and Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

2.1.1.4 Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of Axitinib in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.

2.1.1.5 Information available or pending regarding possible genetic alterations that can explain the patient's pheochromocytoma/paraganglioma (mutations in succinate dehydrogenase-B (SDHB), SDHV or Von Hippel-Lindau (VHL) genes)

2.1.1.6 Last dose of chemotherapy or experimental therapy more than 4 weeks (6 weeks in the case of nitrosourea) prior to enrollment date; 2 weeks if the last therapy was received as part of a phase 0 or exploratory Investigational New Drug (IND) trial. Last surgery more than 4 weeks prior to enrollment, to allow for wound healing. Core biopsies or fine needle aspiration (FNA) will not require any waiting period

2.1.1.7 Last radiotherapy treatment greater than or equal to 4 weeks prior to starting treatment with this protocol and there must be sites of measurable disease that did not receive radiation

2.1.1.8 Prior therapeutic Metaiodobenzylguanidine (MIBG) is allowed

2.1.1.9 Organ and marrow function as defined below:

2.1.1.10 Total bilirubin less than or equal to 1.5 x upper limit of normal (ULN) (upper limit of normal), unless the patient meets the criteria for Gilbert's Syndrome. The upper limit value for bilirubin for subjects with Gilbert's Syndrome is less than 3 mg/dl.

Note: A diagnosis of Gilbert's disease will be made in the presence of (1) unconjugated hyperbilirubinemia noted on several occasions; (2) normal results from complete blood count (CBC) count, reticulocyte count, and blood smear; (3) normal liver function test results; and (4) an absence of other disease processes that can explain the unconjugated hyperbilirubinemia.

2.1.1.11 Aspartate aminotransferase (AST) less than or equal to 2.5 x ULN, alanine aminotransferase (ALT) less than or equal to 2.5 x ULN

2.1.1.12 Amylase and lipase equal to, or less than, the institutional ULN.

2.1.1.13 Creatinine clearance greater than or equal to 40 ml/min (estimated or measured creatinine clearance) or serum creatinine less than or equal to 1.6 mg/dl

2.1.1.14 Random urine protein < 20 mg/dL. If greater than or equal to 20 mg/dL then a 24-hour urine protein collection will be performed to accurately demonstrate that the 24-hour total is <1000 mg, the level acceptable for enrollment on study

2.1.1.15 Absolute neutrophil count greater than or equal to 500/mm(3)

2.1.1.16 Platelet count greater than or equal to 50,000/ mm(3)

2.1.1.17 Ability to understand and sign an informed consent document.

2.1.1.18 Ability and willingness to follow the guidelines of the clinical protocol including visits to National Institute of Child Health and Human Development (NICHD) and National Cancer Institute (NCI), Bethesda, Maryland for treatment and follow up visits.

2.1.1.19 Because the effects of chemotherapy on the developing human fetus are potentially harmful, women of childbearing potential and men who participate in the study must agree to use adequate contraception (hormonal or barrier methods) before, during the study and for a period of 3 months after the last dose of chemotherapy.

EXCLUSION CRITERIA

2.1.2.1 Patients with pheochromocytoma/paraganglioma tumors potentially curable by surgical excision alone as determined by the Principal Investigator in discussions with the surgical consultants

2.1.2.2 Patients who have large abdominal masses impinging on bowel or pulmonary masses with encroached vessels and a potential to bleed will be considered on case by case basis after careful consultation with multiple disciplines such as radiologists and surgeons with main intent being patient safety.

2.1.2.3 Unstable hypertension defined as a systolic blood pressure >150 mm Hg or diastolic pressure > 90 mmHg despite optimal medical management.

2.1.2.4 Untreated brain metastases (or local treatment of brain metastases within the last 6 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic adverse events.

2.1.2.5 Pregnancy, due to the possible adverse effects on the developing fetus.

2.1.2.6 Lactating women who are breast-feeding due to the possibility of transmitting axitinib to the child.

2.1.2.7 The presence of a second malignancy, other than squamous cell carcinoma of the skin or in situ cervical cancer because it will complicate the primary objective of the study. Cancer survivors who have been free of disease for at least two years can be enrolled in this study.

2.1.2.8 Patients with evidence of a bleeding diathesis

2.1.2.9 Patients must not have received prior therapy with a tyrosine kinase inhibitor (TKI). Prior TKI usage in pheochromocytoma affects the same pathway as axitinib.

2.1.2.10 Gastrointestinal abnormalities including:

* Inability to take oral medications
* Requirement for intravenous alimentation
* Prior surgical procedure affecting absorption including total gastric resection
* Treatment for active peptic ulcer disease in the past 6 months
* Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy
* Malabsorption syndrome

2.1.2.11 Current use or anticipated need for treatment with drugs that are known potent Cytochrome P450 3A4 (CYP3A4) inhibitors (i.e., grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, and delavirdine).

2.1.2.12 Current use or anticipated need for treatment with drugs that are known CYP3A4 or Cytochrome P450 1A2, (CYP1A2) inducers (i.e., carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).

2.1.2.13 Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devices or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.

2.1.2.14 Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.

2.1.2.15 Any of the following within 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and within 6 months before study drug administration for deep vein thrombosis or pulmonary embolism.

2.1.2.16 Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10-19 (Actual); Primary Completion 2015-06-29 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein PP, Black HR. A simplified diagnostic approach to pheochromocytoma. A review of the literature and report of one institution's experience. Medicine (Baltimore). 1991 Jan;70(1):46-66. doi: 10.1097/00005792-199101000-00004. PMID 1988766
- [Background] Pacak K, Linehan WM, Eisenhofer G, Walther MM, Goldstein DS. Recent advances in genetics, diagnosis, localization, and treatment of pheochromocytoma. Ann Intern Med. 2001 Feb 20;134(4):315-29. doi: 10.7326/0003-4819-134-4-200102200-00016. PMID 11182843
- [Background] Bravo EL. Pheochromocytoma: new concepts and future trends. Kidney Int. 1991 Sep;40(3):544-56. doi: 10.1038/ki.1991.244. No abstract available. PMID 1787652
- [Derived] Burotto M, Edgerly M, Poruchynsky M, Velarde M, Wilkerson J, Kotz H, Bates S, Balasubramaniam S, Fojo T. Phase II Clinical Trial of Ixabepilone in Metastatic Cervical Carcinoma. Oncologist. 2015 Jul;20(7):725-6. doi: 10.1634/theoncologist.2015-0104. Epub 2015 Jun 3. PMID 26040622
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0001.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/Arm 1-Axitinib
Started | 14
Completed | 7
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Progressed/Removed from treatment | 1
Not completed — Study closing at site | 1
Not completed — Adverse Event | 1
Not completed — Refused further treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | 1/Arm 1-Axitinib
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response (Partial Response + Complete Response)
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or no-target) must have reduction in short axis to <10 mm. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Patients were assessed every 12 weeks (+/- week) up to 40.6 months
Population: 2/14 participants were not evaluated for this outcome measure. Current Investigator inherited this trial when the original investigator left the National Institutes of Health (NIH). The reason participants were not evaluated is unknown.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1-Axitinib
Number analyzed (Participants) | 12
Participants
  Confirmed Partial Response | 5
  Complete Response | 0
  Stable Disease | 5
  Progressive Disease | 2

2. Secondary Outcome: Progression - Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first. Disease progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: time from start of treatment to time of progression or death, up to 5 years and 9 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1/Arm 1-Axitinib
Number analyzed (Participants) | 12
months | 7.7 [3.3 to 16.8]

3. Secondary Outcome: Change in Vascular Endothelial Growth Factor Receptors (VEGFR) in Blood in Metastatic, Recurrent or Primary Unresectable Pheochromocytoma/Paraganglioma
Description: The measurement of VEGFR in blood will be performed using a semi-quantitative immunohistochemistry assay.
Time Frame: up to 3 years
Population: Blood samples were collected on a subset of participants, but assays were never performed on any of the samples and therefore no data for the Outcome Measures were collected.
Arm/Group | 1/Arm 1-Axitinib
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacogenomics Analyses
Description: Measuring genetic alterations.
Time Frame: up to 3 years
Population: as for outcome 3
Arm/Group | 1/Arm 1-Axitinib
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Plasma Levels of Axitinib
Description: Pharmacokinetic analysis will be done to determine drug levels in blood.
Time Frame: Baseline and 3 years
Population: as for outcome 3
Arm/Group | 1/Arm 1-Axitinib
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 54 months and 29 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Arm 1-Axitinib
Number analyzed (Participants) | 14
Participants | 14

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 54 months and 29 days.
Arm/Group | 1/Arm 1-Axitinib
All-Cause Mortality (participants affected / at risk) | 9/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm 1-Axitinib (N=14)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Arm 1-Axitinib (N=14)
Abdominal pain (Gastrointestinal disorders) | 6 (16)
Activated partial thromboplastin time prolonged (Investigations) | 2 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (7)
Alkaline phosphatase increased (Investigations) | 7 (11)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 10 (30)
Anorexia (Metabolism and nutrition disorders) | 5 (10)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Creatinine increased (Investigations) | 5 (15)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (2)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (28)
Dizziness (Nervous system disorders) | 7 (11)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Duodenal infection (Infections and infestations) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Edema limbs (General disorders) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Facial pain (General disorders) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Fatigue (General disorders) | 13 (33)
Fever (General disorders) | 5 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (9)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (13)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (13)
Hypertension (Vascular disorders) | 14 (345)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (20)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 7 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (18)
Hypotension (Vascular disorders) | 5 (11)
Hypothyroidism (Endocrine disorders) | 5 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lipase increased (Investigations) | 2 (3)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 12 (42)
Lymphocyte count increased (Investigations) | 1 (1)
Malaise (General disorders) | 2 (5)
Mitral valve disease (Cardiac disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 7 (44)
Multi-organ failure (General disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (3)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (25)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Neutrophil count decreased (Investigations) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Otitis externa (Ear and labyrinth disorders) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 1 (3)
Pain (General disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (12)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (12)
Palpitations (Cardiac disorders) | 5 (9)
Paresthesia (Nervous system disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Personality change (Psychiatric disorders) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2)
Platelet count decreased (Investigations) | 6 (16)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (10)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary valve disease (Cardiac disorders) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, cystocele (Renal and urinary disorders) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (4)
Sinusitis (Infections and infestations) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Tricuspid valve disease (Cardiac disorders) | 1 (2)
Upper respiratory infection (Infections and infestations) | 6 (9)
Urinary tract infection (Infections and infestations) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (2)
Vaginal stricture (Reproductive system and breast disorders) | 1 (1)
Vaginismus (Reproductive system and breast disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (14)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 5 (10)
White blood cell decreased (Investigations) | 6 (13)
Renal and urinary disorders - Other, hydronephrosis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT01967576/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT01967576/ICF_001.pdf